CLINICAL TRIAL: NCT02062229
Title: Oxidative Stress, Vitamin E and Lipidomics in Seminal Fluid as Potential Link to Infertility
Brief Title: Oxidative Stress and Lipidomics in Male Infertility
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Civic Hospital, Italy (Other)
Responsible Party: Principal Investigator, Luigi Iuliano, M.D., University of Roma La Sapienza
Other Study IDs: IULIANO_Rago
Record Dates: First submitted 2014-02-07; First posted 2014-02-13 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Male Infertility
Keywords: oxidative stress; oxysterols; fatty acids; seminal fluid
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Collection of male seminal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Halthy controls: Subjects not affected by any disease and with normal seminal fluid characteristics
- Oligospermia: Infertile subjects with oligospermia
- Varicocele: Infertile subjects with varicocele
- Asthenospermia: Infertile subjects with asthenospermia

SUMMARY:
Infertility is a common problem, affecting perhaps one couple in six, the majority of whom now seek medical care. It is becoming a social challenge because it is responsible for personal and interpersonal discomfort and anxiety. A major obstacle to meaningful study of the epidemiology of male infertility is the difficulty in accurate diagnosis of the presence or absence of a problem. Traditionally, the diagnosis of male infertility is facilitated by the conventional assessment of the semen profile - constructed according to recognized guidelines (i.e. WHO) and including pH, cell count and motility - but no specific biomarkers are available.

We sought to determine the oxysterol and fatty acid lipidome with the ai of finding a lipid biomarker useful for the diagnosis of male infertility.

DETAILED DESCRIPTION:
Subjects referring to an outpatient infertility laboratory will be enrolled in the study. A complete clinical record is collected as well as a sperm and a fasting blood sample. Patients are stratified according to current guidelines focusing on sperm and anatomical characteristics. Sperm characteristics will be studied on fresh samples immediately after collection; blood samples will be centrifuged and plasma stored at -80°C until analysis that include routine glucose and lipid profile by commercial kits. Vitamin E (alpha- and gamma-tocopherol), oxysterols profiling, and fatty acids profiling is analyzed by state of the art gas chromatography-mass spectrometry (GC/MS) using isotope dilution methods.

ELIGIBILITY:
Inclusion Criteria:

* clinically healthy subjects and clinical healthy subjects with infertility

Exclusion Criteria:

* subjects with endocrine, cardiovascular, metabolic, inflammatory and neurologic diseases or cancer
* subjects taking medicines and/or supplements

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects referring to an infertility center
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Oxysterol profiling in seminal fluid | 1 day
  Oxysterol profiling will be assessed in seminal fluid by state of the art GC/MS

SECONDARY OUTCOMES:
Fatty acids lipidomics | 1 day
  Profiling of fatty acids in seminal fluid will be assessed by GC/MS

OTHER OUTCOMES:
Vitamin E concentration in seminal fluid | 1 day
  the two main vitamin isoforms, alpha- and gamma-tocopherol, will be measured by GC/MS

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Rago, M.D., Principal Investigator — Civic Hospital; Luigi Iuliano, M.D., Study Director — University of Roma La Sapienza
Locations (1):
- Civic Hospital, Fertility Unit, Latina, Italy

REFERENCES:
- [Derived] Zerbinati C, Caponecchia L, Rago R, Leoncini E, Bottaccioli AG, Ciacciarelli M, Pacelli A, Salacone P, Sebastianelli A, Pastore A, Palleschi G, Boccia S, Carbone A, Iuliano L. Fatty acids profiling reveals potential candidate markers of semen quality. Andrology. 2016 Nov;4(6):1094-1101. doi: 10.1111/andr.12236. Epub 2016 Sep 27. PMID 27673576